CLINICAL TRIAL: NCT06985264
Title: Effects of Orbicularis Oculi and Fat Excision on Dry Eye in Upper Blepharoplasty: A Comparative Evaluation
Brief Title: Dry Eye in Upper Eyelid Surgery: Muscle Versus Fat Removal
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Furkan Çiftci, MD, Mersin Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEŞEH
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Eye Disorders
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1) Patients who are currently undergoing Upper Eyelid Blepharoplasty 2) Patients between the ages o (Experimental)
  Interventions: Procedure: Upper Eyelid Blepharoplasty surgery

INTERVENTIONS:
Procedure: Upper Eyelid Blepharoplasty surgery — Orbicularis oculi excision

SUMMARY:
The aim of this study is to compare the effects of two different surgical techniques (Orbicularis Oculi excision and Orbicularis Oculi + Fat excision) applied in upper blepharoplasty surgery on dry eye and to evaluate the effects of these techniques on ocular surface health. 142 patients (71 patients in each group) who met the inclusion and exclusion criteria between 01.05.2025 and 31.12.2025 in Mersin City Education and Research Hospital Eye Diseases Clinic will be included in this study. This study is a prospective, survey study and aims to evaluate the effects of two different surgical techniques (Orbicularis Oculi excision only and Orbicularis Oculi + Fat excision) applied in upper blepharoplasty surgery on postoperative dry eye symptoms. The study will be conducted on patients who are currently scheduled for upper blepharoplasty surgery and no additional surgical procedures or interventions will be applied to the patients. Data collection will be done by a survey study and retrospective recording of routine clinical examinations.

The collected data will be used to analyze the differences in dry eye parameters between the two surgical techniques. OSDI scores, BUT times, Oxford staining degrees, Schirmer test results and visual acuity values will be compared at pre- and postoperative time points. Differences between groups will be analyzed by one-tailed independent samples t-test and p<0.05 will be considered significant. These analyses will be performed to determine the effect of surgical techniques on dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are currently undergoing Upper Eyelid Blepharoplasty
2. Patients between the ages of 18-80
3. Patients with a 6-month postoperative follow-up
4. Patients without a preoperative dry eye diagnosis
5. Patients who have not had previous eyelid surgery
6. Those who signed the Informed Consent Form/Written Consent Form
7. Patients with complete treatment and follow-up files

Exclusion Criteria:

1. Being under 18 and over 80
2. Having a history of previous eyelid surgery
3. Diabetics
4. Having diseases that cause dry eyes such as Sjögren, Systemic Lupus Erythematosus
5. Having dry eye disease before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Preoperative, postoperative 1st month, 3rd month and 6th month Ocular Surface Disease Index (OSDI) score survey will be conducted.
  The OSDI, which was created by the Outcomes Research Group at Allergan Inc in order to quickly assess the symptoms of ocular irritation in dry eye disease and how they affect functioning related to vision. This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin City Education and Research Hospital, Mersin, Çukurova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to restrictions their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Background] Bottomley A, Jones D, Claassens L. Patient-reported outcomes: assessment and current perspectives of the guidelines of the Food and Drug Administration and the reflection paper of the European Medicines Agency. Eur J Cancer. 2009 Feb;45(3):347-53. doi: 10.1016/j.ejca.2008.09.032. Epub 2008 Nov 14. PMID 19013787
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152